CLINICAL TRIAL: NCT03629028
Title: Single or Double-layer Uterine Closure Techniques Following Cesarean: An Ongoing Debate
Brief Title: Single or Double-layer Uterine Closure Techniques
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Safak Baran Yilmaz (Other)
Responsible Party: Sponsor-Investigator, Safak Baran Yilmaz, Specialist Dr. Şafak YILMAZ BARAN M.D., Baskent University
Organization: Baskent University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KA 18/71
Record Dates: First submitted 2018-08-09; First posted 2018-08-14 (Actual); Results first posted 2020-05-01 (Actual); Last update posted 2020-05-01 (Actual); Status verified 2020-04

CONDITIONS: Uterine Scar; Cesarean Section Complications; Cesarean Section; Dehiscence
Keywords: cesarean section, niche, isthmocele, uterine closure

STUDY DESIGN:
Intervention Model Description: Prospective Randomised Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single Layer (Active Comparator): Diagnostic Test: Niche Presence in 6 to 9 months Diagnostic Test: Niche Measurements (depth of niche, the length of niche, the width of the niche in the transverse plane) Diagnostic Test: Residual myometrium thickness Diagnostic Test: Adjacent myometrium thickness Symptoms: postmenstrual bleeding/dysmenorrhea
  Interventions: Diagnostic Test: Residual myometrium thickness; Diagnostic Test: Niche Presence; Diagnostic Test: Adjacent myometrium thickness; Diagnostic Test: Niche Measurements (depth of niche, width of niche, length of niche)
- Double Layer (Active Comparator): Diagnostic Test: Niche Presence in 6 to 9 months Diagnostic Test: Niche Measurements (depth of niche, the length of niche, the width of the niche in the transverse plane) Diagnostic Test: Residual myometrium thickness Diagnostic Test: Adjacent myometrium thickness Symptoms: postmenstrual bleeding/dysmenorrhea
  Interventions: Diagnostic Test: Residual myometrium thickness; Diagnostic Test: Niche Presence; Diagnostic Test: Adjacent myometrium thickness; Diagnostic Test: Niche Measurements (depth of niche, width of niche, length of niche)

INTERVENTIONS:
Diagnostic Test: Residual myometrium thickness — The myometrium will be closed by single or double layer during cesarean and residual myometrium thickness will be evaluated in 6 to 9 months by saline infusion sonography.
Diagnostic Test: Niche Presence — The myometrium will be closed by single or double layer during cesarean and niche presence will be evaluated in 6 to 9 months by saline infusion sonography.
Diagnostic Test: Adjacent myometrium thickness — The myometrium will be closed by single or double layer during cesarean and adjacent myometrium thickness will be evaluated in 6 to 9 months by saline infusion sonography.
Diagnostic Test: Niche Measurements (depth of niche, width of niche, length of niche) — The myometrium will be closed by single or double layer during cesarean and three dimensional niche measurements will be evaluated in 6 to 9 months by saline infusion sonography.

SUMMARY:
There are different surgical techniques of uterine closure during cesarean. A growing data has suggested that the closure technique has an effect on uterine scar healing. Residual myometrium thickness and uterine scar defect (niche) development seems to be related to the single or double layer closure of uterus. In that study, investigators will search for the effect of single or double layer closure of uterus during cesarean on the uterine scar defect.

DETAILED DESCRIPTION:
Study design and participants This study will be assessed cesarean delivery (CD) patients who will admit to the Obstetrics and Gynecology Clinic of the Başkent University Adana Dr. Turgut Noyan Research and Application Center between July 2018 and September 2019. Specifically, participants will be singleton pregnancy patients between 18-45 years of age who will be in gestational weeks 24-41 and had not previously received any uterine operations such as CS or myomectomy. Patients with multiple pregnancies and/or chronic inflammatory diseases such as systemic lupus erythematosus, rheumatoid arthritis, and insulin-dependent diabetes mellitus will be excluded. All patients who meet the inclusion criteria will be randomized into two treatment groups (i.e., single- or double-layer closures).

This study was approved by Başkent University Institutional Review Board and Ethics Committee (Project no= KA18-71, Approval Date= 7/27/2018), and supported by Başkent University Research Fund. Patients who will agree to participate in the study will be informed about the purpose of the study before their operations, and each provided signed written consent.

Participants will be also assessed for maternal age, gravidity, parity, body mass index, smoking status, diabetes mellitus, hypertensive diseases of pregnancy, and medical history. Regardless of whether they had contractions before surgery, this study also will be determined patient CD indications, levels of cervical dilatation, and how CD will be established (i.e., elective or emergent).

Randomization and masking A table of random numbers is used as a simple randomization method for placing participants into the two treatment groups. The Research Randomizer website (https://www.randomizer.org/) was used to create this table. Before the intervention, the next envelope among a previously prepared, sealed, and the number-ordered stack will be opened by a nurse for each procedure.

Surgery technique Six operators will perform CD operations. Access to the abdomen will be achieved via Pfannenstiel incision, while the Kerr incision technique will be applied to the uterus for all patients. Patients in the single-layer group will be received uterus closures with locking, while patients in the double-layer group will be received uterus closures with locking in the first layer, but without locking and using the Lambert style in the second layer. The decidua will be deliberately excluded during all suturations. A synthetic absorbable suture material (Vicryl 1.0, Ethicon, Somerville, NJ, USA) will be used during all uterus closures, with corner stitches that will be applied to all patients. Additional suture usages and numbers will be reported only in cases of bleeding. Both uterine closure and whole operation times will be recorded by the respective operating room technicians. Finally, intravenous prophylactic antibiotics (2 g cefazolin sodium) and uterotonic medications (10 IU oxytocin) will be routinely applied during all CD procedures.

Follow-up Postoperative follow-ups will be completed in March 2020. All participants will be called after delivery and will be invited to complete sixth-month evaluations. However, participants who will experience post-CD pregnancies or uterine surgeries will be excluded. All remaining participants will be examined at six to nine months period after CD for niche presence in the scar region, niche measurements, scar shape, distance between niche and the external cervical os and residual myometrium thickness (RMT), and adjacent myometrium thicknesses (AMT). The distance between the niche and external os should be measured parallel to the top of the main niche, from the most distal niche point to external os. These examinations will be conducted by two experienced sonographers who will be blinded to clinical information regarding the closure technique. Procedures will be specifically completed using a 4-10 MHz transducer (E8C-RS micro convex endocavity probe, Voluson S6, GE, Milwaukee, US), ultrasonography, and through the saline infusion sonohysterography (SIS) method. The cervix will be first cleaned with povidone iodine while the patient will be on the gynecological examination table prior to ultrasonography. The SIS process then will be progressed toward the inside of the endometrial cavity by passing from the cervical os with an intrauterine insemination cannula (intrauterine insemination catheter, Wallace Artificial Insemination Catheter, Smiths Medical International Ltd., Ashford, Kent, UK). A sterile saline solution will be applied to sufficiently distend the cavity, while ultrasonography will be conducted via transvaginal probe. At this time, the presence of a hypoechogenic area with a depth of 2mm or deeper in the CD scar region within the endometrial cavity will be accepted as a niche. Niche dimensions will be determined via 3-axis measurements for depth, length, and width. Niche shape, distance to the external cervical os, RMT, and AMT will be evaluated. During these follow-ups, patients will be also asked about their menstruation processes and any experiences of cervical pain, menstruation pain, postmenstrual bleeding (PMB) in the form of spotting, and other abnormal bleeding patterns. Those who will experience bleeding for two days or more in the form of spotting after menstruation will be defined as PMB. Participants who will use intrauterine devices after CD and/or those who could not tolerate speculum application will be examined via transvaginal ultrasonography (TV USG).

Outcomes Primary outcomes will be considered niche presence and measurements, while secondary outcomes will be considered RMT, AMT, healing ratio, postmenstrual spotting, and dysmenorrhea.

Statistical analyses The sample size was calculated based on a study by Di Spiezio Sardo et al. (2017) titled Risk of Cesarean Scar Defect Following Single- vs Double-Layer Uterine Closure: Systematic Review and Meta-Analysis of Randomized Controlled Trials. Their study revealed niche formation rates for single- and double-layer closure types of 25% and 43%, respectively. Based on tools available at the Power and Sample Size website (http://powerandsamplesize.com/Calculators), the needed sample size was calculated at 141 for each treatment group with 90% power and 0.05 alpha error.

All data were statistically analyzed using the IBM SPSS 21.0 software. Categorical measurements will be presented as frequencies and percentages, while continuous measurements will be summarized as means and standard deviations (median and range when needed). Distributions will be checked and the student's t-test was will be used for variables meeting the parametric test assumptions when comparing the continuous measurements based on groups, while the Mann Whitney U test will be used for those that will not meet the parametric test assumptions. Finally, chi-square or Fisher's test statistics will be used to compare categorical variables. Statistical significance is set to 0.05 for all tests.

ELIGIBILITY:
Inclusion Criteria:

* Primary cesarean, singleton pregnancy,

Exclusion Criteria:

* Multiple pregnancy, History of any uterine surgery, wound healing diseases (insulin dependent diabetes mellitus, rheumatoid arthritis, systemic lupus erythematous, inflammatory bowel disease)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only women who underwent cesarean section
Enrollment: 282 (Actual)
Dates: Start 2018-08-18 (Actual); Primary Completion 2018-08-18 (Actual); Study Completion 2020-03-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Şafak YILMAZ BARAN, M.D., Principal Investigator — Baskent University Department of Obstetrics and Gynecology
Locations (1):
- Baskent University Adana Seyhan Uygulama Hastanesi, Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Di Spiezio Sardo A, Saccone G, McCurdy R, Bujold E, Bifulco G, Berghella V. Risk of Cesarean scar defect following single- vs double-layer uterine closure: systematic review and meta-analysis of randomized controlled trials. Ultrasound Obstet Gynecol. 2017 Nov;50(5):578-583. doi: 10.1002/uog.17401. Epub 2017 Oct 9. PMID 28070914

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Layer: Age:18-45 Years,Only women who underwent cesarean section Inclusion Criteria:Primary cesarean, singleton pregnancy, Exclusion Criteria:Multiple pregnancy, History of any uterine surgery, wound healing diseases (insulin dependent diabetes mellitus, rheumatoid arthritis, systemic lupus erythematous, inflammatory bowel disease) Uterus will be sutured in locked single layer during cesarean Diagnostic Test: Total myometrium thickness, Residual myometrium thickness, Niche Presence and Measurements in 3D will be evaluated in 6th months by saline infusion sonography.
- Double Layer: Age:18-45 Years,Only women who underwent cesarean section Inclusion Criteria:Primary cesarean, singleton pregnancy, Exclusion Criteria:Multiple pregnancy, History of any uterine surgery, wound healing diseases (insulin dependent diabetes mellitus, rheumatoid arthritis, systemic lupus erythematous, inflammatory bowel disease) Uterus will be sutured in double layer during cesareanDiagnostic Test: Total myometrium thickness, Residual myometrium thickness, Niche Presence and Measurements in 3D will be evaluated in 6th months by saline infusion sonography.
Period: Overall Study
Arm/Group | Single Layer | Double Layer
Started (18/08/2018) | 141 | 141
Completed | 109 | 116
Not Completed | 32 | 25
Not completed — Lost to Follow-up | 26 | 23
Not completed — Pregnancy | 4 | 2
Not completed — intolerance to examination | 2 | 0

BASELINE CHARACTERISTICS:
Population: same ethnic origin, 18-45 age, who underwent first cesarean operation
Groups:
- Single Layer: uterus will be sutured by single layer
- Double Layer: uterus will be sutured by double layer
- Total: Total of all reporting groups
Arm/Group | Single Layer | Double Layer | Total
Number analyzed (Participants) | 109 | 116 | 225
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.8 (4.1) | 30.8 (5.1) | 30.3 (4.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 109 | 116 | 225
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 109 | 116 | 225
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 28.9 (4.2) | 29.8 (4.6) | 29.3 (4.4)
Gestational age at delivery [Mean (Standard Deviation); unit: weeks] | 38 (2) | 38.1 (2.1) | 38.1 (2)
birth weight [Mean (Standard Deviation); unit: g] | 3191.5 (570) | 3261.4 (633) | 3227.3 (602.8)
Tobacco use [Count of Participants; unit: Participants] | 5 | 4 | 9
Diabetes mellitus [Count of Participants; unit: Participants] | 6 | 9 | 15
Hypertension in pregnancy [Count of Participants; unit: Participants] | 10 | 9 | 19
History of infertility [Count of Participants; unit: Participants] | 22 | 25 | 47
Nulliparity [Count of Participants; unit: Participants] | 103 | 105 | 208
Emergent cesarean section [Count of Participants; unit: Participants] | 30 | 35 | 65
Contractions before labor [Count of Participants; unit: Participants] | 29 | 34 | 63
≥4 cm cervical dilatation [Count of Participants; unit: Participants] | 11 | 14 | 25
Need for additional suture [Count of Participants; unit: Participants] | 64 | 66 | 130
Duration of uterine closure [Median (Full Range); unit: min] | 3.5 [1 to 9] | 6.15 [1.5 to 20] | 5.2 [1 to 20]
Operation time [Median (Full Range); unit: min] | 25 [15 to 45] | 30 [20 to 50] | 27 [15 to 50]
Duration of labor [Median (Full Range); unit: hour] | 1 [1 to 18] | 1 [1 to 20] | 1 [1 to 20]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Niche Visualized by Saline Infusion Sonography
Description: The presence of niche in incision line visualized by saline infusion sonography
Time Frame: 6 to 9 months
Measure: Count of Participants; unit: Participants
Groups:
- Single Layer; Double Layer: niche presence
Arm/Group | Single Layer | Double Layer
Number analyzed (Participants) | 109 | 116
Participants
  number and percentage of niche by saline infusion | 40 | 53
  the presence of niche by tv ultrasound | 25 | 23
Statistical Analysis 1: Comparison: Single Layer vs Double Layer; The sample size was calculated based on the study of Sardo et al. The website http://powerandsamplesize.com/Calculators was used. As a result of the sample size calculation with 90% power and 0.05 alpha error, it was planned to include 141 patients in each group; Test type: Non-Inferiority — Data compared to meta-analysis conducted in Sardo et al., 2017; p = 0.05, Chi-squared; Chi-squared or Fisher's test statistic was used to compare the categorical variables

2. Primary Outcome: Median Depth of Niche
Description: with saline infusion sonohysterography
Time Frame: 6-9 months
Measure: Median (Full Range); unit: mm
Groups:
- Single Layer: single layer median depth of niche
- Double Layer: double layer median depth of niche
Arm/Group | Single Layer | Double Layer
Number analyzed (Participants) | 109 | 116
mm | 1.7 [0 to 8.4] | 2.4 [0 to 6.3]

3. Primary Outcome: Median Length of Niche
Description: by saline infusion sonohysterography
Time Frame: 6-9 months
Population: of the 225 partipicants included the study
Measure: Median (Full Range); unit: mm
Groups:
- Single Layer; Double Layer: median length niche
Arm/Group | Single Layer | Double Layer
Number analyzed (Participants) | 109 | 116
mm | 3.5 [0 to 6.7] | 3.8 [0 to 9.3]

4. Primary Outcome: Median Width of Niche in Transverse Plane
Description: median width of niche in transverse plane by saline infusion sonohysterograhpy
Time Frame: 6-9 months
Population: of the 225 participants included the study
Measure: Median (Full Range); unit: mm
Groups:
- Single Layer; Double Layer: median niche width in transverse plane
Arm/Group | Single Layer | Double Layer
Number analyzed (Participants) | 109 | 116
mm | 2.8 [0 to 7.4] | 4 [0 to 10.1]

5. Secondary Outcome: Residual Myometrium Thickness - 6 to 9 Months
Description: The residual myometrium thickness in incision line measured by saline infusion sonography
Time Frame: 6 to 9 months
Measure: Median (Full Range); unit: mm
Groups:
- Single Layer; Double Layer: Residual myometrium thickness
Arm/Group | Single Layer | Double Layer
Number analyzed (Participants) | 109 | 116
mm | 9.6 [3.7 to 21] | 9.4 [3 to 23]

6. Secondary Outcome: Adjacent Myometrium Thickness
Description: Adjacent myometrium thickness out of incision line measured by saline infusion sonography
Time Frame: 6 to 9 months
Measure: Median (Full Range); unit: mm
Groups:
- Single Layer; Double Layer: Adjacent myometrium thickness
Arm/Group | Single Layer | Double Layer
Number analyzed (Participants) | 109 | 116
mm | 12.1 [6.8 to 22.6] | 12 [4.9 to 23]

ADVERSE EVENTS:
Time Frame: 6 months
Description: no serious adverse event occured
Groups:
- Single Layer-; Double Layer: Presence of niche, niche measurements, measurement of residual/ adjacent myometrium thickness
Arm/Group | Single Layer- | Double Layer
All-Cause Mortality (participants affected / at risk) | 0/109 | 0/116
Serious Adverse Events (participants affected / at risk) | 0/109 | 0/116
Other Adverse Events (participants affected / at risk) | 1/109 | 0/116
OTHER ADVERSE EVENTS (reported when occurring in more than 1.1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Layer- (N=109) | Double Layer (N=116)
pregnancy occurred after cesarean (Pregnancy, puerperium and perinatal conditions) | 1 (4) | NA (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-07-27): https://cdn.clinicaltrials.gov/large-docs/28/NCT03629028/Prot_SAP_ICF_000.pdf